CLINICAL TRIAL: NCT00593996
Title: Evaluation of Potential Vitamin D Effects on Muscle: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-1224
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-05

CONDITIONS: Dysphagia; Fecal Incontinence; Urinary Incontinence
MeSH Terms: conditions — Deglutition Disorders; Fecal Incontinence; Urinary Incontinence | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Placebo Comparator): oral placebo 3 times weekly
  Interventions: Other: Ergocalciferol (vitamin D2)

INTERVENTIONS:
Other: Ergocalciferol (vitamin D2) — 50,000 IU 3 times weekly for 4 weeks

SUMMARY:
People who do not have adequate amounts of vitamin D develop weakness of leg and arm muscles. This study will determine if vitamin D supplementation benefits muscle functions important for swallowing, bladder and bowel function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present for evaluation to the UW Geriatric clinic including Dr. Pryzbelski's subspecialty, or Osteoporosis clinics
* Age 70 years or older
* Cognitively intact, as determined by the attending physicians at above mentioned clinics

Exclusion Criteria:

* History of, on ongoing, renal failure
* History of liver failure
* Known malabsorption
* Known disorders of parathyroid function, hyper/hypocalcemia, or other abnormalities of calcium or phosphate metabolism
* Known history of vitamin D intoxication or granulomatous disease
* active seizure disorder
* Pain associated with temporomandibular joint (TMJ)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-07; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
change in lingual strength and perceived swallow function | 4 weeks

SECONDARY OUTCOMES:
change in perceived bowel and bladder function | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Principal Investigator — Univ. of Wisconsin - Institute on Aging
Locations (1):
- UW Osteoporosis Clinical Research Program, Madison, Wisconsin, United States